CLINICAL TRIAL: NCT01794754
Title: May Occupational Therapy Delay the Need for Surgery in Carpometacarpal Osteoarthritis: A Randomised Controlled Trial.
Brief Title: Occupational Therapy and Surgery in Carpometacarpal Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Resource Center for Rehabilitation in Rheumatology (Other)
Collaborators: St. Olavs Hospital (Other); Haukeland University Hospital (Other); Haugesund Rheumatism Hospital (Other)
Responsible Party: Principal Investigator, Ingvild Kjeken, Senior researcher, National Resource Center for Rehabilitation in Rheumatology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012/2265-3
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis in the Carpometacarpal (CMC) Joint
Keywords: Hand osteoarthritis; CMC1-joint; surgery; occupational therapy; hand exercises; assistive devices; orthoses
MeSH Terms: conditions — Capillary Malformations, Congenital, 1 | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Care as usual
  Interventions: Other: Care as usual
- Occupational therapy (Experimental): Occupational therapy
  Interventions: Other: Occupational therapy

INTERVENTIONS:
Other: Care as usual
  Arms: Control
Other: Occupational therapy — Occupational therapy in the waiting period before surgery. Occupational therapy comprises orthoses for the CMC-joint, hand exercises, and use of alternative working methods and assistive devices. The participants are encouraged to perform hand exercises three times a week for the first 12 weeks, and to use orthosis as much as possible, both during daytime (day orthosis) and night time (night orthosis).
  Arms: Occupational therapy

SUMMARY:
The purpose of the study is to investigate if occupational therapy may delay or prevent the need for surgery in patients with carpometacarpal(CMC) osteoarthritis (OA) who are scheduled for surgery in the CMC-joint.

Our study hypothesis is that compared to participants in the intervention group, significantly more participants in the control group have received CMC-surgery after two years.

DETAILED DESCRIPTION:
Hand osteoarthritis (OA) is one of the most prevalent musculoskeletal diseases in an adult population, and approximately 68% of people between the ages of 71 and 80 years have radiographic OA in the carpometacarpal (CMC) joint.

Currently, there is no cure for hand OA. However, several studies have demonstrated that hand exercises and CMC-orthoses may reduce pain and improve grip strength, and in a recent study, assistive devices improved activity performance and satisfaction with performance in people with hand-OA. Still, most people do not receive any such treatment, but those with severe CMC-OA are often referred for surgery in this joint. The effect of occupational therapy to prevent or delay need for surgery CMC-OA has been investigated in a small study with 33 participants, but randomised controlled trails (RCT) of good quality are needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CMC-OA who are referred for review for the need for surgery in the CMC joint.

Exclusion Criteria:

* Persons with cognitive dysfunction
* Persons who do not understand the Norwegian language
* Persons with other diseases or injuries that may negatively impact hand function

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Number of participants in each group who have received surgery. | Two years

SECONDARY OUTCOMES:
Hand Pain at rest and in activity | Two years
  Measured on Numeric Rating Scales, 0 - 10.
Number of painful hand joints. | Two years
  Examination.
Joint mobility in 2-5 finger. | Two years
  Flexion deficit in millimetre.
Thumb flexion. | Two years
  Goniometer
Thumb abduction. | Two years
  Pollexograph.
Grip strength. | Two years
  Grip-It, measured in Newton)
Pinch strength | Two years
  Grip-It, measured in Newton
Activity performance. | Two years
  MAP-Hand - a patient reported outcome/questionnaire.
Hand and shoulder function | Two Years
  Quick-Dash, a patient reported outcome/questionnaire
Satisfaction with care. | Two years
  On Numeric Rating Scales, 0 - 10.
Health related quality of life. | Two years
  EQ5D, a patient reported outcome/questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Tore K Kvien, PhD, Study Director — Research director, Diakonhjemmet Hospital
Locations (4):
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Haugesund Rheumatism Hospital, Haugesund
  - National resource center for rehabilitation in rheumatology, Oslo
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kjeken I, Eide RE, Klokkeide A, Matre KH, Olsen M, Mowinckel P, Andreassen O, Darre S, Nossum R. Does occupational therapy reduce the need for surgery in carpometacarpal osteoarthritis? Protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2016 Nov 15;17(1):473. doi: 10.1186/s12891-016-1321-3. PMID 27842579
- [Background] Kjeken I, Eide RE, Klokkeide A, Matre KH, Olsen M, Mowinckel P, Andreassen O, Darre S, Nossum R. Erratum to: Does occupational therapy reduce the need for surgery in carpometacarpal osteoarthritis? Protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2017 Feb 6;18(1):68. doi: 10.1186/s12891-017-1433-4. No abstract available. PMID 28166750
- [Derived] Tveter AT, Kleven L, Osteras N, Nossum R, Eide REM, Klokkeide A, Matre KH, Olsen M, Kjeken I. Is multimodal occupational therapy in addition to usual care cost-effective in people with thumb carpometacarpal osteoarthritis? A cost-utility analysis of a randomised controlled trial. BMJ Open. 2023 Jun 23;13(6):e063103. doi: 10.1136/bmjopen-2022-063103. PMID 37355263
- [Derived] Tveter AT, Osteras N, Nossum R, Eide REM, Klokkeide A, Matre KH, Olsen M, Kjeken I. Short-Term Effects of Occupational Therapy on Hand Function and Pain in Patients With Carpometacarpal Osteoarthritis: Secondary Analyses From a Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2022 Jun;74(6):955-964. doi: 10.1002/acr.24543. Epub 2022 Apr 5. PMID 33338325
- See also: Link to free full text of protocol in BMC musculoskeletal disorders — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5109819/
- See also: Link to free full text of erratum protocol in BMC musculoskeletal disorders — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5109819/